CLINICAL TRIAL: NCT01950468
Title: Evaluation of the Diagnostic Efficacy and Safety of [123I]NAV5001 as an Imaging Agent to Aid in the Diagnosis of Parkinsonian Syndromes
Brief Title: A Cross-Over, Multi-Center Trial to Evaluate the Diagnostic Efficacy and Safety of [123I]NAV5001 as an Imaging Agent to Aid in the Diagnosis of Parkinsonian Syndromes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The entire drug development program for this molecule was sold to another company.
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV5-02
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Syndrome
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — ioflupane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAV5001 (Experimental)
  Interventions: Drug: NAV5001
- DaTscan (Active Comparator)
  Interventions: Drug: DaTscan

INTERVENTIONS:
Drug: NAV5001 — A single intravenous dose of 8.0 ± 1.0 mCi
  Arms: NAV5001
Drug: DaTscan — A single intravenous dose of 3 to 5 mCi
  Arms: DaTscan

SUMMARY:
This is a phase 3, open-label, multiple-center, randomized cross-over study to assess the safety and efficacy of [123I]NAV5001 SPECT imaging in aiding in the differentiaion of parkinsonian syndromes from non-parkinsonian tremor.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent before the initiation of any study related procedures and continues to give willing consent for participation
* Age ≥ 40 years
* Have had upper extremity tremor for < 3 years duration, regardless of presumed diagnosis or etiology
* Have a UPDRS part III score upon entry of ≤ 16

Exclusion Criteria:

* Any clinically significant or unstable physical or psychological illness based on medical history or physical examination at screening, as determined by the investigator
* Structural brain abnormality affecting the entire brain (e.g., normal pressure hydrocephalus) or the striatum (e.g., local tumor or stroke)
* Any clinically significant abnormal laboratory results obtained at screening and as determined by the investigator
* Any clinically significant abnormal electrocardiogram (ECG) results obtained at screening and as determined by the investigator
* Any history of drug, narcotic, or alcohol abuse within 2 years before the date of informed consent, as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, Fourth Edition, revised (DSM-IV-TR [American Psychiatric Association, 1994])
* Positive urine drug screen for opiates, cocaine, or amphetamines at screening
* Positive pregnancy test before imaging
* Participation in an investigational drug or device clinical trial within 30 days before the date of informed consent
* Previous scan with any DAT imaging agent (e.g. [123I]NAV5001, Altropane, DaTscan, DOPASCAN)
* Any exposure to radiopharmaceuticals within 30 days before the date of informed consent
* Breast-feeding
* Inability to lie supine for 1 hour
* Any thyroid disease other than adequately treated hypothyroidism
* Known sensitivity or allergy to iodine or iodine containing products
* Treatment within the 30 days before the date of imaging with amoxapine, amphetamine, benztropine, bupropion, buspirone, cocaine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, selegiline, and sertraline, paroxetine, or citalopram.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of Parkinson' Syndrome based on the Movement Disorder Specialist Consensus Panel | One Year
The incidence of positve [123I]NAV5001 SPECT brain scans | Baseline
The incidence of Parkinson' Syndrome based on the on-site neurologist assessment | Baseline

SECONDARY OUTCOMES:
The incidence of Parkinson' Syndrome based on the on-site neurologist assessment at 6 months | 6 months
The incidence of Parkinson' Syndrome based on the on-site neurologist assessment at 1 year | 1 Year
Incidence of adverse events post baseline | 1 year

OTHER OUTCOMES:
The incidence of positve DaTscan SPECT brain scans | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Reininger, M.D. Ph.D., Study Director — Navidea Biopharmaceuticals
Locations (2):
- United States (2):
  - Xenoscience, Inc., Phoenix, Arizona
  - Compass Research, Orlando, Florida